CLINICAL TRIAL: NCT03168308
Title: Sugammadex Versus Neostigmine for Reversal of Rocuronium-induced Neuromuscular Blockade: A Study of Thoracic Surgical Patients
Brief Title: Sugammadex vs. Neostigmine for Neuromuscular Blockade Reversal in Thoracic Surgical Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Tiffany B Moon, Assistant Professor, Director of Resident Research, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STU 032017-030
Record Dates: First submitted 2017-05-23; First posted 2017-05-30 (Actual); Results first posted 2020-02-19 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: Neuromuscular Blockade
MeSH Terms: interventions — Sugammadex; Glycopyrrolate

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Neostigmine & Glycopyrrolate (Active Comparator): Patients randomized to receive Neostigmine w/ Glycopyrrolate
  Interventions: Drug: Neostigmine w/ Glycopyrrolate
- Sugammadex (Active Comparator): Patients randomized to receive Sugammadex
  Interventions: Drug: Sugammadex

INTERVENTIONS:
Drug: Sugammadex — Sugammadex 2 mg/kg
  Arms: Sugammadex
Drug: Neostigmine w/ Glycopyrrolate — Neostigmine 50 mcg/kg, maximum 5 mg Glycopyrrolate, 8 mcg/kg, maximum 1 mg
  Arms: Neostigmine & Glycopyrrolate

SUMMARY:
This prospective, randomized, double blinded study is intended to enroll a total of 92 patients undergoing thoracic surgery with general endotracheal anesthesia at Parkland Hospital. Patients will be randomized to receive either neostigmine or sugammadex for reversal of neuromuscular blockade. Merck, Inc. will supply the sugammadex through an agreement with Parkland Investigational Drug Services. Neostigmine is readily available for anesthesiologists to use and is the current standard of care for reversal of neuromuscular blockade. A standardized anesthetic protocol that is usual and customary for the type of operation the patient is having will be provided to the anesthesia teams of enrolled subjects. The remainder of the anesthetic care of the subject will not deviate from the standard of care. The surgeon, anesthesia team, postoperative recovery nurse, and research assistant will be blinded as to which reversal drug the patient receives. The only individual that will know to which drug the patient has been randomized will be the pharmacist who draws up the medication(s). A blinded research assistant will record postoperative outcomes and the patient will be followed 90 minutes postoperatively for any adverse events.

DETAILED DESCRIPTION:
Screening and Informed Consent:

A member of the research team will use a screening form to look for surgical patients that meet all of the inclusion and exclusion criteria. He/she will approach potential subjects during pre-anesthesia evaluation clinic (PAEC). Patients who are unable to be consented in PAEC will be approached in the preoperative area and the study will be explained in detail in a private room. Patients will be informed that they will receive no compensation for participating in the study and there will be no adverse consequences if they choose not to participate. If the subjects agree to participate, informed written consent will be obtained prior to any study procedures and this document will be sent to pmhresearchparticipants@phhs.org, for inclusion in the patient's medical record, per Parkland regulations. The study duration is from the start of anesthesia to 90 minutes postoperatively.

Anesthesia Protocol:

The anesthesia team that will be caring for the subject during surgery will be given the protocol for the study, which standardizes the general anesthetic technique. All patients will receive 0.6 mg/kg of rocuronium for neuromuscular paralysis during induction. Additional rocuronium will be given in 0.15 mg/kg increments to keep the patient at a neuromuscular depth of 1 twitch throughout the surgery. All patients will have the depth of neuromuscular block monitored at the non-dominant ulnar nerve at 60 mA with a TOF Watch accelerometer device, which provides real time feedback of the strength of contraction and graphically displays the relevant ratios.

Maintenance of anesthesia will be with sevoflurane in 70% oxygen, titrated to keep the bispectral index (BIS) between 40-60. All patients will have a forced air warming device (e.g., Bair Hugger, 3M, Maplewood, MN) used to maintain normothermia throughout the surgery. Subjects will be randomized to receive blinded study drug: either neostigmine or sugammadex for reversal of neuromuscular blockade, which will be administered intravenously at the beginning of skin closure. The anesthesia team will be blinded. The blinded study drug (reversal agent(s)) will be prepared into a 10 mL syringe by a pharmacist in Investigational Drug Service (IDS) Pharmacy and labeled in a blinded fashion as "sugammadex or neostigmine/glycopyrrolate." Any volume of blinded study drug (reversal agent(s)) that is less than 10 mL will be supplemented with 0.9% normal saline solution, preservation-free so that all syringes contain a volume of 10 mL and appear identical in order to preserve blinding. Any patient with clinical signs of inadequate reversal or failure of recovery of neuromuscular function [TOFR < 0.2] at 20 min after reversal will receive a rescue dose of sugammadex. The remaining aspects of the anesthetic will be standardized and not differ from the standard of care and will be similar for all patients.

Randomization & Dosing:

Patients will be randomized to one of two groups for reversal of neuromuscular paralysis:

1. Group 1- neostigmine (NEO group)

   1. Neostigmine 50 mcg/kg, maximum 5 mg
   2. Glycopyrrolate, 8 mcg/kg, maximum 1 mg
2. Group 2- sugammadex (SUG group). a. Sugammadex 2 mg/kg

The research coordinator will make randomization envelopes by using a random number generator. These envelopes will be provided to IDS Pharmacy before any subjects are screened and later only as needed to replenish supply. The words 'neostigmine/glycopyrrolate' or 'sugammadex' will be printed on a piece of paper and placed in an opaque manila envelope that bears a unique subject number (#). Upon receiving the physician order for the subject, the IDS Pharmacist will randomize the subject to a treatment group by opening the randomization envelope bearing the subject # corresponding to the subject # written on the physician order.

The Investigator or Co-Investigator will write the patient's total body weight (TBW) on the physician order so that the pharmacist can perform necessary dose calculations and draw up the appropriate intravenous dose of the blinded study drug (reversal agent(s)): sugammadex OR neostigmine/glycopyrrolate. After the blinded study drug syringe is prepared, a pharmacist or pharmacy technician will deliver the syringe to the operating room to the anesthesia provider, who will sign for receipt of the study drug syringe.

Blinding/Un-blinding:

The patient, all medical providers (surgeons, anesthesia faculty, anesthesia residents, certified registered nurse anesthetists, nurses), and the postoperative evaluator will be blinded as to what reversal agent (sugammadex versus neostigmine/glycopyrrolate) the patient receives. A member of the research team that is not involved in the direct care or assessment of the patient will provide the randomization envelopes to IDS Pharmacy. IDS Pharmacy staff will be the only un-blinded personnel.

In emergency scenarios where un-blinding becomes necessary (e.g., anaphylaxis), the Principal Investigator or Co-Investigators may call the IDS Pharmacy to ascertain which specific medication(s) was dispensed. A detailed log of patient enrollments, randomization assignments and drug accountability will be kept in Investigational Drug Service (IDS) Pharmacy, which has controlled security access.

Calculation of Key Times:

The time that the reversal agent (sugammadex versus neostigmine) is given will be marked as 'Reversal Time', and times to last stitch, extubation, and out of OR will be ascertained from the electronic medical record (EMR) (i.e., Epic Systems, Verona, WI). A trained research assistant will assess the degree of neuromuscular function the patient has in the early postoperative period. Adequate reversal will be defined as a train of four ratio (TOFR) ≥ 0.9. Anything less than 0.9 will be defined as residual paralysis or inadequate reversal.

Postoperative Recovery Assessment:

A blinded, trained research assistant will observe and record all parameters during the early postoperative period. All episodes of hypoxia will be recorded and any use of supplemental oxygen will be recorded. A standard O2 weaning protocol will be used in the PACU. All vital signs will be extracted from the EMR. Any drugs given will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years old
* Undergoing non-emergent thoracic surgery
* ASA physical status classification 2 to 4
* Willing and able to consent in English or Spanish
* No personal history of neuromuscular disease

Exclusion Criteria:

* Age less than 18 or older than 80
* Patient does not speak English or Spanish
* Planned postoperative intubation or ICU admission
* Allergy to sugammadex, neostigmine, glycopyrrolate, or rocuronium
* Family or personal history of malignant hyperthermia
* Patient refusal
* Monitored anesthesia care (MAC) or regional anesthesia planned
* Pregnant or nursing women
* "Stat" (emergent) cases
* Estimated creatinine clearance <30 mL/min
* Pre-existing muscle weakness of any etiology
* Patients on toremifene (a selective estrogen receptor modulator)
* Women on oral contraceptives who do not wish to use a non-hormonal method of contraception for 7 days following surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2017-09-26 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany Moon, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Parkland Health & Hospital System, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Neostigmine & Glycopyrrolate | Sugammadex
Started | 48 | 44
Completed | 48 | 44
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Neostigmine & Glycopyrrolate | Sugammadex | Total
Number analyzed (Participants) | 48 | 44 | 92
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 48 | 44 | 92
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.9 (13.8) | 53.1 (14.4) | 51.1 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 22 | 48
  Male | 22 | 22 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 20 | 41
  Not Hispanic or Latino | 27 | 24 | 51
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 48 | 44 | 92

OUTCOME MEASURES:

1. Primary Outcome: Number of Hypoxic Episodes
Description: Hypoxia was defined as an episode of peripheral oxygen saturation (SpO2) <94% on ≤2 L/min of oxygen by nasal cannula, or a SpO2 <98% on ≥2 L/min of oxygen, or postoperative SpO2 of ≥5% reduction compared to preoperative values.
Time Frame: Through patient's stay in the early postoperative period, approximately 1-2 hours.
Measure: Median (Inter-Quartile Range); unit: episode(s)
Arm/Group | Neostigmine & Glycopyrrolate | Sugammadex
Number analyzed (Participants) | 48 | 44
episode(s) | 1 [0 to 2.2] | 0 [0 to 1]

2. Secondary Outcome: Time to Complete Reversal of Neuromuscular Blockade
Description: The time from the administration of the blinded reversal syringe until complete reversal of neuromuscular blockade (train of four ratio ≥0.9).
Time Frame: From time of reversal to complete reversal of neuromuscular blockade (train of four ratio ≥0.9), approximately 1 hour
Measure: Mean (Inter-Quartile Range); unit: minutes
Arm/Group | Neostigmine & Glycopyrrolate | Sugammadex
Number analyzed (Participants) | 48 | 44
minutes | 40 [15 to 53] | 10 [5 to 15]

3. Secondary Outcome: Number of Participants Who Needed Rescue Sugammadex After Initial Reversal of Neuromuscular Blockade
Description: To determine if reversal with sugammadex versus neostigmine requires an additional dose of sugammadex rescue after initial reversal of neuromuscular blockade.
Time Frame: From time of reversal to 80 minutes after arrival in the post-anesthesia care unit, approximately 1-2 hours.
Measure: Count of Participants; unit: Participants
Arm/Group | Neostigmine & Glycopyrrolate | Sugammadex
Number analyzed (Participants) | 48 | 44
Participants | 5 | 0

ADVERSE EVENTS:
Time Frame: Monitored for 24 hours after surgery end time.
Arm/Group | Neostigmine & Glycopyrrolate | Sugammadex
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/44
Serious Adverse Events (participants affected / at risk) | 5/48 | 0/44
Other Adverse Events (participants affected / at risk) | 0/48 | 0/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neostigmine & Glycopyrrolate (N=48) | Sugammadex (N=44)
Reintubation (Surgical and medical procedures) | 1 (1) | 0 (0)
Critical respiratory or circulatory events (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Symptoms of residual neuromuscular blockade (Injury, poisoning and procedural complications) | 5 (5) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-07): https://cdn.clinicaltrials.gov/large-docs/08/NCT03168308/Prot_SAP_002.pdf